CLINICAL TRIAL: NCT03527498
Title: A Randomized Clinical Trial of Infant Treadmill for Long-term Neurodevelopmental Evaluation of Neonatal Encephalopathy
Brief Title: Evaluation of Long-term Neurodevelopment in Neonatal Encephalopathy by Infant Treadmill
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The other study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai 6F+ Early intervention center for high risk preterm infants (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHFudanU_NNICU8
Record Dates: First submitted 2018-02-22; First posted 2018-05-17 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Periventricular Leukomalacia; Intraventricular Hemorrhage; Bilirubin Encephalopathy; Kernicterus; Hypoglycemia, Neonatal; Cerebral Infarction
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Leukomalacia, Periventricular; Kernicterus; Hypoglycemia; Cerebral Infarction

STUDY DESIGN:
Intervention Model Description: All subjects were divided into two groups: intervention group A (treadmill intervention + routine physical rehabilitation therapy) and positive control group (receiving routine physical rehabilitation therapy only).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Baby treadmill + physical rehabilitation training
  Interventions: Device: Baby treadmill; Behavioral: Physical rehabilitation training
- positive control group (Active Comparator): Physical rehabilitation training only
  Interventions: Behavioral: Physical rehabilitation training

INTERVENTIONS:
Device: Baby treadmill — The newborns who received treadmill intervention were stimulated by running 3 times a week for a total of 10 minutes each time (complete in 5 cycles, 2 minutes per cycle, 2 minutes after the completion of one cycle and rest for 2 minutes to start the next cycle). Until the completion and completion of the five cycles). During the remaining four days of each week, other physical rehabilitation training is carried out by the rehabilitator in accordance with the established rehabilitation plan. The stimulation of running lasted from 3 months of corrected gestational age to being able to walk alone for 3 steps or to correct for 18 months.
  Arms: intervention group
Behavioral: Physical rehabilitation training — Suitable for general physical rehabilitation training of all infants with cerebral palsy.

SUMMARY:
There is no international application of infant running stimulation system to evaluate the brain injury in children with various stages of nerve and motor development in a large sample of studies. The study of neonatal brain injury is only limited to intraventricular hemorrhage(IVH),periventricular leukomalacia(PVL), Down's syndrome(DS), premature birth of these four conditions, and the number of samples in the single digits, there is no representative of the disease population. Therefore, from the newborn to the infant development of the critical period, the investigator will refer to the previous treadmill parameters set on the research results, optimize the application of neonatal treadmill. The study hypothesized that neonatal treadmill stimulation with brain-injured children could improve his / her staggered gait characteristics and long-term nerve development through large sample data. It is important to preserve and analyze the gait characteristics and the changes of nerve development in every stage of growth and development of neonates with brain injury so as to provide clinical evidence for rehabilitation intervention. It is of great significance to judge whether this technique can be used in the early stage of brain injury in neonates.

DETAILED DESCRIPTION:
There is no international application of infant running stimulation system to evaluate the brain injury in children with various stages of nerve and motor development in a large sample of studies. The study of neonatal brain injury is only limited to intraventricular hemorrhage(IVH),periventricular leukomalacia(PVL), Down's syndrome(DS), premature birth of these four conditions, and the number of samples in the single digits, there is no representative of the disease population. Therefore, from the newborn to the infant development of the critical period, the investigators will refer to the previous treadmill parameters set on the research results, optimize the application of neonatal treadmill. The study hypothesized that neonatal treadmill stimulation with brain-injured children could improve his / her staggered gait characteristics and long-term nerve development through large sample data. It is important to preserve and analyze the gait characteristics and the changes of nerve development in every stage of growth and development of neonates with brain injury so as to provide clinical evidence for rehabilitation intervention. It is of great significance to judge whether this technique can be used in the early stage of brain injury in neonates.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age < 33 weeks;
2. Correction of gestational age < 3 months;
3. It has been diagnosed as hypoxic-ischemic encephalopathy, periventricular intraventricular hemorrhage, periventricular leukomalacia, bilirubin encephalopathy, persistent hypoglycemia and cerebral infarction.
4. There was no other therapeutic intervention before entering the study;
5. Informed consent is signed by the family.

Exclusion Criteria:

This study is excluded from the study provided that one of the following conditions is met:

1. Brain injury caused by central or peripheral infection (cerebrospinal fluid positive / torch test positive / three major conventional culture positive);
2. Brain damage caused by convulsion;
3. Metabolic brain damage caused by genetic defects;
4. Suffering from known severe congenital malformations;
5. Definite head trauma during labor or postpartum;
6. Peripheral neuromuscular disease or abnormal skeletal system.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
score from Bayley Scales of Infant and Toddler Development testing | The length of time from birth to the corrected age of 18 months
  These scores are largely used for screening, helping to identify the need for further observation and intervention, as infants who score very low are at risk for future developmental problems.
fractional anisotropy(FA) | The length of time from birth to the corrected age of 18 months
  a variable from Diffusion Tensor Image（DTI）sequence of MRI
the value of Amplitude of Low Frequency Fluctuation(ALFF) | The length of time from birth to the corrected age of 18 months
  a variable from resting-blood oxygenation level dependent（BOLD）sequence of MRI

SECONDARY OUTCOMES:
Alberta Infant Motor Development Assessment | The length of time from birth to the corrected age of 18 months
  Neurodevelopmental evaluation scale
Peabody motor development scale | The length of time from birth to the corrected age of 18 months
  The Peabody Developmental Motor Scales (PDMS) is composed of six subtests that measure interrelated abilities in early motor development. It was designed to assess gross and fine motor skills in children from birth through five years of age. Reflexes (Re), Stationary (St), Locomotion (Lo) , Object Manipulation (Ob), Grasping (Gr), Visual-Motor Integration (Vi). All of the PDMS-2 subtests contribute to a Total Motor Quotient (TMQ).
Gross Motor Function Measure Scale | The length of time from birth to the corrected age of 18 months
  There is a 4-point scoring system for each item on the GMFM. Specific descriptors for scoring items are detailed in the administration and scoring guidelines. The GMFM-66 requires a user-friendly computer programme called the Gross Motor Ability Estimator, or GMAE, to enter individual item scores and convert them to an interval level total score.
the value of regional homogeneity (ReHo) | Corrected age of 18 months
  a variable from resting-blood oxygenation level dependent（BOLD）sequence of MRI
mean diffusion(MD) | The length of time from birth to the corrected age of 18 months
  a variable from Diffusion Tensor Image（DTI） sequence of MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasudevan EV, Patrick SK, Yang JF. Gait Transitions in Human Infants: Coping with Extremes of Treadmill Speed. PLoS One. 2016 Feb 1;11(2):e0148124. doi: 10.1371/journal.pone.0148124. eCollection 2016. PMID 26828941
- [Background] Teulier C, Lee DK, Ulrich BD. Early gait development in human infants: Plasticity and clinical applications. Dev Psychobiol. 2015 May;57(4):447-58. doi: 10.1002/dev.21291. Epub 2015 Mar 18. PMID 25782975
- [Background] Siekerman K, Barbu-Roth M, Anderson DI, Donnelly A, Goffinet F, Teulier C. Treadmill stimulation improves newborn stepping. Dev Psychobiol. 2015 Mar;57(2):247-54. doi: 10.1002/dev.21270. Epub 2015 Feb 2. PMID 25644966
- [Background] de Klerk CC, Johnson MH, Heyes CM, Southgate V. Baby steps: investigating the development of perceptual-motor couplings in infancy. Dev Sci. 2015 Mar;18(2):270-80. doi: 10.1111/desc.12226. Epub 2014 Aug 13. PMID 25123212
- [Background] Madhavan S, Campbell SK, Campise-Luther R, Gaebler-Spira D, Zawacki L, Clark A, Boynewicz K, Kale D, Bulanda M, Yu J, Sui Y, Zhou XJ. Correlation between fractional anisotropy and motor outcomes in one-year-old infants with periventricular brain injury. J Magn Reson Imaging. 2014 Apr;39(4):949-57. doi: 10.1002/jmri.24256. Epub 2013 Oct 17. PMID 24136687
- [Background] Angulo-Barroso RM, Tiernan C, Chen LC, Valentin-Gudiol M, Ulrich D. Treadmill training in moderate risk preterm infants promotes stepping quality--results of a small randomised controlled trial. Res Dev Disabil. 2013 Nov;34(11):3629-38. doi: 10.1016/j.ridd.2013.07.037. Epub 2013 Sep 4. PMID 24012586